CLINICAL TRIAL: NCT03256864
Title: A Six-month, Prospective, Single-center, Pilot Study Determining the Pharmacokinetics and Effectiveness of Twice-daily Tacolimus and Everolimus Regimen Convert to Once-daily Tacrolimus and Everolimus Regimen in Liver Transplant Patients
Brief Title: Twice-daily Tacrolimus and Everolimus Convert to Once-daily Tacrolimus and Everolimus in Liver Transplant Recipient
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Wei-Chen Lee, Chief of transplanet center, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CRAD001HTW02T
Record Dates: First submitted 2016-02-01; First posted 2017-08-22 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Liver Transplantation
MeSH Terms: interventions — Tacrolimus; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tacrolimus and Everolimus BID (Experimental): TAC BID (C0 2.5-5 ng/mL) EVR BID (1.0 mg BID targeted to C0 3-8 ng/mL)
  Other Names:
  * Prograf
  * Advagraf
  * Zortress
  * Certican
  Interventions: Drug: Tacrolimus and Everolimus
- Tacrolimus and Everolimus QD (Experimental): TAC QD (C0 2.5-5 ng/mL) EVR QD (2.0 mg QD targeted to C0 3-8 ng/mL)
  Other Names:
  * Prograf
  * Advagraf
  * Zortress
  * Certican
  Interventions: Drug: Tacrolimus and Everolimus

INTERVENTIONS:
Drug: Tacrolimus and Everolimus — In the TAC and EVR BID arm, everolimus will be initiated at a dose of 1.0 mg BID within 24 h of randomization with the dose adjusted from day 5 onward to maintain trough (C0) concentration in the range 3-8 ng/mL. Tacrolimus will be initiated at a dose of 0.15 mg/kg BID and then taper to 0.10 mg/kg BID to maintain trough (C0) concentration in the range 2.5-5 ng/mL.
  In the TAC and EVR QD arm, everolimus will be initiated at a dose of 2.0 mg QD within 24 h of randomization with the dose adjusted from day 5 onward to maintain trough (C0) concentration in the range 3-8 ng/mL. Tacrolimus will be initiated at a dose of 0.1-0.2 mg/kg/day QD to maintain trough (C0) concentration in the range 2.5-5 ng/mL.
  Other Names: Prograf; Advagraf; Zortress; Certican

SUMMARY:
It has been identified that nonadherence to immunosuppressant regimen may cause long-term graft failure and death in solid organ transplant recipients. Therefore, simplification of the immunosuppression regimen by reducing daily dosing frequency may improve long-term outcome. The investigators will examine pharmacokinetics and safety profiles of stable liver transplant recipients receiving twice-daily TAC with EVR (BID) regimen and then being converted to once-daily TAC with EVR (QD) regimen over a 6-month study period post-conversion.

DETAILED DESCRIPTION:
Randomized trial of everolimus (EVR) with reduced tacrolimus (TAC) regimen after liver transplantation has shown similar incidence of composite efficacy failure rate to a standard tacrolimus regimen, but with superior renal function for up to three years. Recent studies have demonstrated comparable efficacy and safety profiles in liver transplant recipients receiving tacrolimus once-daily (QD) and tacrolimus twice-daily (BID) regimens. In kidney transplantation, once daily everolimus (QD) regimen has shown its safety and effectiveness. It has been identified that nonadherence to immunosuppressant regimen may cause long-term graft failure and death in solid organ transplant recipients. Therefore, simplification of the immunosuppression regimen (e.g. TAC with EVR) by reducing daily dosing frequency may improve long-term outcome. However, little is known about the effectiveness and safety of combined TAC and EVR once-daily (QD) regimen in liver transplant recipients. The investigator will examine pharmacokinetics and safety profiles of stable liver transplant recipients receiving twice-daily TAC with EVR (BID) regimen and then being converted to once-daily TAC with EVR (QD) regimen over a 6-month study period post-conversion.

ELIGIBILITY:
Key inclusion criteria

Stable liver transplant recipients are eligible for inclusion in this study and have to fulfill all of the following criteria:

1. Liver Transplant Recipients have received liver transplantations for at least 6+1 months prior to enrollment
2. Liver Transplant Recipients have no acute rejection episodes within 3 months prior to the enrollment and are clinically stable
3. Liver Transplant Recipients have been treated with twice-daily regimen of tacrolimus(TAC) plus everolimus(EVR) and TAC and EVR trough levels have stayed within targeted ranges for at least 6 weeks prior to enrollment
4. Provide written informed consent prior to inclusion.
5. Liver transplant recipients who are 18-65 years of age of a primary liver transplant
6. Allograft functioning at an acceptable level as defined by the AST, ALT, Total Bilirubin levels ≤3 times ULN prior to enrollment.
7. Abbreviated MDRD eGFR ≥ 30 mL/min/1.73m2. Key exclusion criteria

Patients fulfilling any of the following criteria are not eligible for inclusion in this study:

1. Patients who are recipients of multiple solid organ or islet cell tissue transplants, or have previously received an organ or tissue transplant. Patients who have a combined liver-kidney transplant.
2. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
3. Existence of any surgical, medical or mental conditions, other than the current transplantation, which, in the opinion of the investigator, might interfere with the objectives of the study.
4. Pregnant or nursing (lactating) women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-01; Primary Completion 2019-06-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
To evaluate pharmacokinetic profile of everolimus and tacrolimus in liver transplant recipients on AUC (area under the curve) | 6 month
  Area under the plasma concentration versus time curve (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: WeiChen Lee, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided